CLINICAL TRIAL: NCT00637468
Title: Multizenterstudie Der European Assessment Group for Lysis in the Eye (EAGLE) Zur Behandlung Des Zentralarterienverschlusses (ZAV): Lysetherapie Versus Konservative Therapie
Brief Title: EAGLE - Multicenter Study of the European Assessment Group for Lysis in the Eye
Acronym: EAGLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to results of conditional power analysis performed at the first interim analysis and due to observed spectrum of adverse events.
Sponsor: University Hospital Freiburg (Other)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S 020301
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Retinal Artery Occlusion; Fibrinolysis; Visual Acuity; Stroke; Hemodilution
MeSH Terms: conditions — Retinal Artery Occlusion; Stroke | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Local intra-arterial fibrinolysis (LIF)
  Interventions: Drug: Intravenous injection of heparin; Procedure: Local intra-arterial fibrinolysis
- 2 (Active Comparator): Conservative standard therapy
  Interventions: Drug: Intravenous injection of heparin; Drug: Intravenous injection of acetazolamide; Procedure: Globe massage; Drug: Topical use of beta-blocker; Drug: Isovolaemic haemodilution; Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Intravenous injection of heparin
Drug: Intravenous injection of acetazolamide
  Arms: 2
Procedure: Local intra-arterial fibrinolysis
  Arms: 1
Procedure: Globe massage
  Arms: 2
Drug: Topical use of beta-blocker
  Arms: 2
Drug: Isovolaemic haemodilution
  Arms: 2
Drug: Acetylsalicylic acid
  Arms: 2

SUMMARY:
The aim of the EAGLE Study is to compare the efficacy of conservative medical treatment and local intraarterial fibrinolysis in patients with central retinal artery occlusion and to evaluate benefit and risk for the patient of both therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subtotal central retinal artery occlusion or central retinal artery occlusion with choroidal hypoperfusion not lasting longer than 20h
* Patients aged from 18 years to 75 years (in case of pre-existing blindness of other eye also older than 75 years)
* Informed consent of the patient

Exclusion Criteria:

* Central retinal artery occlusion lasting longer than 20h
* Eye diseases, namely branch retinal artery occlusion, cilioretinal arteries supplying the macula, combined arterial-venous occlusion, proliferative diabetic retinopathy and elevated intraocular pressure (over 30 mmHg)
* Systemic diseases, namely severe general diseases, systemic arterial hypertension (systolic pressure > 200 mmHg), despite medical therapy, acute systemic inflammation (erythrocyte sedimentation rate > 30 mm within the first hour/ C-reactive protein > 1,0 mg/dl), antithrombin-III deficiency in case of thrombocytopenia (< 100000 per ml): pathologic clotting time, acute pancreatitis with elevated pancreas enzymes
* Medical History: heart attack within the last 6 weeks, intracerebral bleeding or neurosurgical operation within the last 4 weeks, therapy with marcumar/warfarin, allergic reaction to contrast agent, haemorrhagic diathesis, aneurysms, inflammatory vascular diseases (e.g., giant cell arteritis, Wegener´s granulomatosis), endocarditis, gastric ulcer
* Patient participation in other studies during the prior 4 weeks
* No willingness and ability of the patient to participate in all follow-up examinations
* Pregnancy
* Written consent not given
* Patient is not mobile (bedridden)
* Other conditions/ circumstances likely to lead to poor treatment adherence (e.g., history of poor compliance, alcohol or drug dependency, no fixed abode)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2002-09

PRIMARY OUTCOMES:
Visual acuity 1 month after therapy in comparison with visual acuity before therapy measured according to ETDRS Scale. | 1 month

SECONDARY OUTCOMES:
Improvement of visual field | 1 month
Effect on retinal circulation | 1 month
Tolerance of therapies and registration of number, form and severity of complications | 1 month
Evaluation of prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schumacher, Professor, Principal Investigator — Department of Neuroradiology, University Medical Center Freiburg
Locations (21):
- Austria (3):
  - Universityhospital Graz, Graz
  - Universityhospital Innsbruck, Innsbruck
  - Allgemeines Krankenhaus Wien, Vienna
- Germany (16):
  - University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universityhospital of RWTH Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Universityhospital Bonn, Bonn
  - UKL Essen, Essen
  - Allgemeines Krankenhaus Hamburg Altona, Hamburg
  - UKE Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universityhospital Homburg/Saar, Homburg/Saar
  - Universityhospital Kiel, Kiel
  - Medizinische Universität zu Lübeck, Lübeck
  - Universityhospital Magdeburg, Magdeburg
  - Universityhospital Mainz, Mainz
  - Universityhospital Marburg, Marburg
  - LMU München, München
  - Universityhospital Würzburg, Würzburg
- Switzerland (2):
  - Universitätsspital Bern, Bern
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Background] Feltgen N, Neubauer A, Jurklies B, Schmoor C, Schmidt D, Wanke J, Maier-Lenz H, Schumacher M; EAGLE-Study Group. Multicenter study of the European Assessment Group for Lysis in the Eye (EAGLE) for the treatment of central retinal artery occlusion: design issues and implications. EAGLE Study report no. 1 : EAGLE Study report no. 1. Graefes Arch Clin Exp Ophthalmol. 2006 Aug;244(8):950-6. doi: 10.1007/s00417-005-0140-2. Epub 2005 Dec 22. PMID 16372192
- [Background] Feltgen N, Reinhard T, Kampik A, Jurklies B, Bruckmann H, Schumacher M. [Lysis therapy vs. conservative therapy: randomised and prospective study on the treatment of acute central retinal artery occlusion (EAGLE study)]. Ophthalmologe. 2006 Oct;103(10):898-900. doi: 10.1007/s00347-006-1429-1. German. PMID 16998653
- [Derived] Pielen A, Pantenburg S, Schmoor C, Schumacher M, Feltgen N, Junker B, Callizo J; EAGLE Study Group. Predictors of prognosis and treatment outcome in central retinal artery occlusion: local intra-arterial fibrinolysis vs. conservative treatment. Neuroradiology. 2015 Oct;57(10):1055-62. doi: 10.1007/s00234-015-1588-3. Epub 2015 Sep 8. PMID 26349479